CLINICAL TRIAL: NCT06682221
Title: EFFECTS of RESISTANCE TRAINING and PROTEIN SUPPLEMENTATION on CARDIORESPIRATORY, METABOLIC, IMMUNOLOGICAL, RENAL and BODY COMPOSITION VARIABLES in ELDERLY INDIVIDUALS
Brief Title: Effects of Resistance Training and Supplementation in Elderly: Cardiorespiratory and Metabolic Variables
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: FundaÃ§Ã£o de Amparo a Pesquisa do Estado de Goias (FAPEG) (Unknown)
Responsible Party: Principal Investigator, Rodolfo de Paula Vieira, BSc., MSc., PhD., Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6.095.284; 202310267000648 (Other Grant/Funding Number: FAPEG)
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Aging; Cardiovascular Health Status; Physical Training; Nutritional Interventions; Respiratory Health; Immunology
Keywords: Elderly; resistance training; metabolism; hemodynamic processes; body composition
MeSH Terms: interventions — Resistance Training; Control Groups

STUDY DESIGN:
Intervention Model Description: The elderly participants will be between 60 and 85 years old and will be randomly assigned to one of four groups, with n = 40 in each group: Control Group (CG; untrained and unsupplemented; n = 40), Supplemented Group (SG; untrained and supplemented; n = 40), Trained Group (TG; trained and unsupplemented; n = 40), and Trained and Supplemented Group (TSG; trained and supplemented; n = 40).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Whey protein supplementation. (Experimental): Protein supplementation will be provided through isolated whey protein, commonly known as whey protein isolate, which was generously donated by the Heroes Science Institute (HSI), as stated in the attached declaration. This whey protein isolate, with a vanilla flavor, is packaged in 25-gram sachets, each providing a total of 20 grams of protein per dose/sachet.
  Interventions: Dietary Supplement: Whey protein supplementation.
- Resistance training (Experimental): The resistance training protocol in the study included seven exercises: high pull, leg extension, leg curl, bicep curl, triceps pushdown, lateral raise, and machine bench press, taking about 60 minutes per session. The first week focused on familiarizing participants with the exercises to ensure proper execution before intensive training began. Training occurred three times a week for 12 weeks, with each exercise performed in 3 sets of 8 to 12 repetitions and rest periods of 1 to 2 minutes. The load was progressively increased by 2% to 10% weekly, based on participants' ability to complete repetitions with full range of motion. Assessments were conducted before training and 24 hours after the final session to evaluate the effects on physical and functional parameters.
  Interventions: Behavioral: Resistance training
- Whey protein supplementation and Resistance training (Sham Comparator): The participants would simultaneously apply both protocols, involving both supplementation and resistance training, to assess the combined effects of these interventions on their health and physical conditioning.
  Interventions: Dietary Supplement: Whey protein supplementation.; Behavioral: Resistance training
- Control (Sham Comparator): The control group will not participate in any of the interventions proposed in the study, meaning it will not receive supplementation or undergo resistance training, serving as a reference to compare the results of the other intervention groups.
  Interventions: Other: Group Control

INTERVENTIONS:
Dietary Supplement: Whey protein supplementation. — Protein supplementation will be provided through isolated whey protein, commonly known as whey protein isolate, which was generously donated by the Heroes Science Institute (HSI), as stated in the attached declaration. This whey protein isolate, with a vanilla flavor, is packaged in 25-gram sachets, each providing a total of 20 grams of protein per dose/sachet.
  Arms: Whey protein supplementation and Resistance training; Whey protein supplementation.
Behavioral: Resistance training — The resistance training protocol in the study included seven exercises: high pull, leg extension, leg curl, bicep curl, triceps pushdown, lateral raise, and machine bench press, taking about 60 minutes per session. The first week focused on familiarizing participants with the exercises to ensure proper execution before intensive training began. Training occurred three times a week for 12 weeks, with each exercise performed in 3 sets of 8 to 12 repetitions and rest periods of 1 to 2 minutes. The load was progressively increased by 2% to 10% weekly, based on participants' ability to complete repetitions with full range of motion. Assessments were conducted before training and 24 hours after the final session to evaluate the effects on physical and functional parameters.
  Arms: Resistance training; Whey protein supplementation and Resistance training
Other: Group Control — The control group will not participate in any of the interventions proposed in the study, meaning it will not receive supplementation or undergo resistance training, serving as a reference to compare the results of the other intervention groups.
  Arms: Control

SUMMARY:
Aging causes losses in strength, lean mass, and cardiovascular health in the elderly due to metabolic changes and alterations in body composition. To investigate whether nutritional interventions and physical training can mitigate these effects, a randomized clinical trial will be conducted at the Evangelical University of Goiás with elderly individuals aged 60 to 85. Participants will be divided into four groups: control, protein supplementation, physical training, and a combination of both. The study will last for 12 months, with evaluations every four months, covering cardiovascular, pulmonary, immunological, renal, muscular, and hematological parameters. The analyses will seek statistical significance, and it is expected that the interventions will significantly improve the participants' health.

DETAILED DESCRIPTION:
The aging process is associated with declines in strength, lean mass (LM), and cardiovascular (CV) and cardiorespiratory (CR) health due to metabolic, hemodynamic, and body composition changes in the elderly. The implications of these changes can potentially be mitigated through nutritional intervention and physical training. To test this hypothesis, a randomized clinical trial will be conducted at the Evangelical University of Goiás (UniEVANGÉLICA), where elderly volunteers (aged 60 to 85) will be randomized (n = 40/group) into control groups (no protein supplementation and no physical training), supplementation group (only protein supplementation), training group (only physical training), and a combined group (physical training + protein supplementation). The supplementation and training protocols will be conducted for 12 months, with evaluations occurring before the protocol begins and every four months thereafter. Numerous cardiovascular, pulmonary, immunological, renal, muscular, and hematological parameters will be assessed. Analyses will be expressed as mean and standard deviation, with a significance level of p≤0.05 for paired t-tests and multiparametric analyses. It is expected that the effects of the resistance training and protein supplementation protocols, together or separately, will significantly improve the described parameters, yielding positive results for the participants.

ELIGIBILITY:
Inclusion Criteria:

- Individuals who volunteer to participate in the study must sign the Informed Consent Form (ICF), be willing to participate in all assessments, and maintain a minimum attendance of 75% in the classes.

Exclusion Criteria:

* Individuals with neurological diseases that prevent them from participating in the assessments and the physical training program will not be eligible.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-16 (Actual); Primary Completion 2024-12-16 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Lung function | Three months
  Pulmonary function will be assessed using a Master Screen spirometer (Jaeger, Germany), employing the forced maneuver in accordance with the standards set by the Brazilian Society of Pneumology and Tisiology. All participants will undergo spirometric testing before and after the administration of a rapid-acting bronchodilator (Salbutamol 400 mcg). The parameters to be evaluated will include Forced Vital Capacity (FVC), Forced Expiratory Volume in the first second (FEV1), the FEV1/FVC ratio, Peak Expiratory Flow (PEF), and Expiratory Flow between 25% and 75% of FVC (FEF25-75).
Pulmonary fibrotic biomarkers | Three months
  The condensed air will be obtained through tidal breathing in a tube called RTube (Respiratory Research, USA), where the volunteer will breathe for a period of 15 minutes. After this period, the condensed air will be collected and stored at -86ºC for the analysis of cytokine levels, growth factors, and anti-fibrotic proteins, as already standardized in our laboratory (Moraes-Ferreira et al., 2022).

CONTACTS AND LOCATIONS:
Locations (1):
- Evangelical University of Goiás - UniEVANGÉLICA, Anápolis, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All data collected and all measurements done will be shared and properly explained to all participants in a private and previously scheduled meeting
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning: 11 December 2024. End: 31 January 2025.
Access Criteria: The principal investigator will have access to IPS and all data through data bank used in the Laboratory of Pulmonary and Exercise Immunology.